CLINICAL TRIAL: NCT03092648
Title: Autologous Bronchial Basal Cells Transplantation for Treatment of Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Regend Therapeutics (Industry); Tongji University (Other)
Responsible Party: Principal Investigator, Guodong HU, Chief Physician, Nanfang Hospital, Southern Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2016-187
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: open, non-random, concurrent control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bronchial basal cells (Experimental)
  Interventions: Biological: Bronchial basal cell
- Control (No Intervention)

INTERVENTIONS:
Biological: Bronchial basal cell — autologous bronchial basal cell transplantation
  Arms: Bronchial basal cells

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a kind of chronic bronchitis or emphysema with characteristics of long-term poor airflow, resulting in chronic pulmonary heart disease, chronic respiratory failure or even death. Anatomically, the pulmonary bronchus structures in COPD patients are damaged and cannot be repaired by recent clinical treatment so far. This study intends to carry out an open, single-armed, phase I/II clinical trial to investigate whether bronchial basal cells can regenerate damaged lung tissue. During the treatment, bronchial basal cells will be isolated from patients' own bronchi and expanded in vitro. After careful characterization, cultured cells will be transplanted autologously into the lesion by fiberoptic bronchoscopy. The safety and efficacy of the treatment will be monitored by measuring the key clinical indicators.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 to 75;
* Diagnosed with COPD according the guideline (a. with symptoms of productive cough, sputum production or shortness of breath; b. with poor airflow as indicated by FEV1<70% predicted value and FEV1/FVC < 0.7 in pulmonary function test; c. with exclusion of other pulmonary disease by CT or blood examination.);
* Clinically stable for more than 4 weeks;
* Tolerant to bronchofiberscope;
* Written informed consent signed.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients positive for syphilis, HIV;
* Patients with malignant tumor;
* Patients with serious significant pulmonary infection and need anti-infection treatment;
* Patients with serious heart disease(NYHA class Ⅲ-Ⅳ);
* Patients with a history of abusing alcohol and illicit drug;
* Patients participated in other clinical trials in the past 3 months;
* Patients assessed as inappropriate to participate in this clinical trial by investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 1-6 months
  One of the indicators for pulmonary function
Forced vital capacity (FVC) | 1-6 months
  One of the indicators for pulmonary function

SECONDARY OUTCOMES:
FEV1/FVC, MMF, MVV and DLCO | 1-6 months
  Other indicators for the pulmonary function
6 minute walk test (6MWT) | 1-6 months
  Indicator to evaluate the exercise function of patients with moderate or severe pulmonary heart diseases
MMRC | 1-6 months
  Indicator to evaluate the level of dyspnea
SGRQ | 1-6 months
  A questionnaire to assess life quality affected by the respiratory problems

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zuo, Ph. D., Study Chair — Regend Therapeutics Co.Ltd
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No